CLINICAL TRIAL: NCT06186778
Title: The Impact of Repeated Colonoscopic Insert Method on the Detection Rate of Adenomas in the Sigmoid Colon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jianning Yao (Other)
Responsible Party: Sponsor-Investigator, Jianning Yao, Deputy Chief Physician, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2023-KY-1332-002
Record Dates: First submitted 2023-11-25; First posted 2024-01-02 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Colorectal Polyp
Keywords: colorectal polyps; colonoscopy; repeat colonoscopy; detection rate; sigmoid colon

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional colonoscopy group (Active Comparator): It starts from the rectum and progresses forward to the cecum, with observations made during withdrawal: from the cecum, ascending colon, transverse colon, descending colon, and sigmoid colon to the rectum.
  Interventions: Procedure: conventional colonoscopy
- secondary colonoscopy group (Experimental): After the routine colonoscopy, a repeat colonoscopy of the sigmoid colon is performed
  Interventions: Procedure: secondary colonoscopy

INTERVENTIONS:
Procedure: secondary colonoscopy — After the routine colonoscopy, a repeat colonoscopy of the sigmoid colon is performed
  Arms: secondary colonoscopy group
Procedure: conventional colonoscopy — It starts from the rectum and progresses forward to the cecum, with observations made during withdrawal: from the cecum, ascending colon, transverse colon, descending colon, and sigmoid colon to the rectum.
  Arms: conventional colonoscopy group

SUMMARY:
Colorectal cancer (CRC) is a malignant tumour originating from the colorectal mucosal epithelium, with rising incidence and mortality rates. Approximately 90% of CRC develops from colorectal polyps, which are considered precancerous lesions of CRC, especially adenomatous polyps. If removed endoscopically during the polyp stage, 70%-90% of CRC can be prevented. However, current colonoscopy examinations have a high miss rate for polyps. Studies have shown that the miss rates for polyps and adenomas after colonoscopy can reach 22%-28% and 12%-26%, respectively.

The "2014 Chinese Guidelines for Early Screening and Endoscopic Diagnosis and Treatment of Colorectal Cancer" mentions that the observation method during colonoscopy starts from the rectum and progresses forward to the cecum, with observations made during withdrawal. However, in actual clinical practice, it is found that single withdrawal observation is not enough, as this examination approach is prone to many missed polyps. The likely reason is that the colon is in a compressed state during withdrawal observation. Single-operator colonoscopy is currently the mainstream insertion method internationally, and the essence of the single-operator technique is "short-axis reductions", meaning that the colonoscope maintains a straight configuration throughout the entire examination. The average adult colon length is about 1.5m, but the distance reached by the colonoscope during the single-operator technique is often between 70-80cm, indicating compression of the colon. In addition, colonic folds become more dense when compressed, making it easier for lesions like polyps to hide within or near folds, leading to misses.

The sigmoid colon, with the most turns in the entire large intestine, is also the part most prone to compression during colonoscopy insertion. Correspondingly, it is also more prone to misses during withdrawal observation. Although some scholars proposed repeating withdrawal to improve lesion detection rates, whether it is performed twice or three times, only compressed colons are observed. In actual clinical work, many polyps can only be found during insertion. The investigators propose performing a second insert specifically for the easily compressed sigmoid colon. During the second insert, the "short-axis reduction" technique should not be used. Instead, the folds should be deliberately advanced into, which helps fully extend the compressed sigmoid colon to shallow or eliminate the folds, allowing observation during advancement to achieve effects beyond multiple withdrawals, finding hidden lesions within or near folds to improve colonoscopy quality. Therefore, to explore whether observing during a second sigmoid colon advancement can further improve the adenoma detection rate to improve colonoscopy quality and reduce interval cancers, the investigators conducted this study.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is a malignant tumour originating from the colorectal mucosal epithelium, with rising incidence and mortality rates. Currently, CRC ranks third in incidence and second in mortality among all cancers worldwide, making it the leading cancer in terms of global incidence and mortality. Approximately 90% of CRC develops from colorectal polyps, which are considered precancerous lesions of CRC, especially adenomatous polyps. If removed endoscopically during the polyp stage, 70%-90% of CRC can be prevented. However, current colonoscopy examinations have a high miss rate for polyps. Studies have shown that the miss rates for polyps and adenomas after colonoscopy can reach 22%-28% and 12%-26%, respectively.

The "2014 Chinese Guidelines for Early Screening and Endoscopic Diagnosis and Treatment of Colorectal Cancer" mentions that the observation method during colonoscopy starts from the rectum and progresses forward to the cecum, with observations made during withdrawal: from the cecum, ascending colon, transverse colon, descending colon, sigmoid colon to the rectum. Current quality control of colonoscopy mainly focuses on controlling withdrawal time exceeding 6 minutes, controlling cecal intubation rate, and ensuring adenoma detection rate, without specific requirements on the observation method. However, in actual clinical practice, it is found that single withdrawal observation is not enough, as this examination approach is prone to many missed polyps. The likely reason is that the colon is in a compressed state during withdrawal observation. Single-operator colonoscopy is currently the mainstream insertion method internationally, and the essence of the single-operator technique is "short-axis reductions", meaning that the colonoscope maintains a straight configuration throughout the entire examination. The average adult colon length is about 1.5m, but the distance reached by the colonoscope during the single-operator technique is often between 70-80cm, indicating compression of the colon. In addition, colonic folds become more dense when compressed, making it easier for lesions like polyps to hide within or near folds, leading to misses. Currently, in the clinical practice of colonoscopy, only withdrawal observation is performed, and only once, on a compressed colon. Many lesions can be easily missed.

The sigmoid colon, with the most turns in the entire large intestine, is also the part most prone to compression during colonoscopy insertion. Correspondingly, it is also more prone to misses during withdrawal observation. Although some scholars proposed repeating withdrawal to improve lesion detection rates, whether it is performed twice or three times, only compressed colons are observed. In actual clinical work, many polyps can only be found during advancement. The investigators propose performing a second advancement specifically for the easily compressed sigmoid colon. During the second advancement, the "short-axis reduction" technique should not be used. Instead, the folds should be deliberately advanced into, which helps fully extend the compressed sigmoid colon to shallow or eliminate the folds, allowing observation during advancement to achieve effects beyond multiple withdrawals, finding hidden lesions within or near folds to improve colonoscopy quality. Therefore, to explore whether observing during a second sigmoid colon advancement can further improve the adenoma detection rate (ADR) to improve colonoscopy quality and reduce interval cancers, the investigators conducted this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent painless colonoscopy at the Gastrointestinal Endoscopy Center of the First Affiliated Hospital of Zhengzhou University and signed the informed consent for the clinical trial;
2. Aged at age 45 and above with BMI >24.

Exclusion Criteria:

1. Patients with contraindications to colonoscopy: patients with acute diverticulitis, patients with known or suspected perforation, patients with severe cardiovascular and cerebrovascular lesions, patients with severe hepatic or renal insufficiency, patients with abdominal aneurysm of large arteries, patients with active hemorrhagic descending colonic lesions, patients with acute radiological colorectal inflammation, patients with advanced carcinomas with pelvic metastases or obvious ascites, patients with severe and extensive intestinal adhesions after abdominal or pelvic surgery;
2. Patients with inflammatory bowel disease, colorectal cancer, familial adenomatous polyposis, Peutz-Jeghers syndrome, abdominal wall hernia, patients with a history of colorectal surgery;
3. Patients with incomplete colonoscopy, i.e., those in whom the endoscopist has failed to successfully cannulate the cecum due to technical difficulties;
4. Patients with poor bowel preparation, i.e., patients with a total score of <6 or any bowel segment of <2 on the Boston Bowel Preparedness Scale score for poor bowel preparation).

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 650 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-05-29 (Actual)

PRIMARY OUTCOMES:
Detection rate of sigmoid colon adenoma | 3 months
  Number of patients with adenomas detected in the sigmoid colon in each group/number of patients examined in each group

SECONDARY OUTCOMES:
Detection rate of sigmoid colon polyps | 3 months
  Number of patients with polyps detected in the sigmoid colon in each group/number of patients examined in each group

CONTACTS AND LOCATIONS:
Locations (1):
- Colonoscopy, Zhengzhou, Henan, China

REFERENCES:
- [Background] Arnold M, Sierra MS, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global patterns and trends in colorectal cancer incidence and mortality. Gut. 2017 Apr;66(4):683-691. doi: 10.1136/gutjnl-2015-310912. Epub 2016 Jan 27. PMID 26818619
- [Background] Shaukat A, Kahi CJ, Burke CA, Rabeneck L, Sauer BG, Rex DK. ACG Clinical Guidelines: Colorectal Cancer Screening 2021. Am J Gastroenterol. 2021 Mar 1;116(3):458-479. doi: 10.14309/ajg.0000000000001122. PMID 33657038
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Song M, Emilsson L, Bozorg SR, Nguyen LH, Joshi AD, Staller K, Nayor J, Chan AT, Ludvigsson JF. Risk of colorectal cancer incidence and mortality after polypectomy: a Swedish record-linkage study. Lancet Gastroenterol Hepatol. 2020 Jun;5(6):537-547. doi: 10.1016/S2468-1253(20)30009-1. Epub 2020 Mar 17. PMID 32192628
- [Background] Zauber AG, Winawer SJ, O'Brien MJ, Lansdorp-Vogelaar I, van Ballegooijen M, Hankey BF, Shi W, Bond JH, Schapiro M, Panish JF, Stewart ET, Waye JD. Colonoscopic polypectomy and long-term prevention of colorectal-cancer deaths. N Engl J Med. 2012 Feb 23;366(8):687-96. doi: 10.1056/NEJMoa1100370. PMID 22356322
- [Background] Zhao S, Wang S, Pan P, Xia T, Chang X, Yang X, Guo L, Meng Q, Yang F, Qian W, Xu Z, Wang Y, Wang Z, Gu L, Wang R, Jia F, Yao J, Li Z, Bai Y. Magnitude, Risk Factors, and Factors Associated With Adenoma Miss Rate of Tandem Colonoscopy: A Systematic Review and Meta-analysis. Gastroenterology. 2019 May;156(6):1661-1674.e11. doi: 10.1053/j.gastro.2019.01.260. Epub 2019 Feb 6. PMID 30738046
- [Background] Martinez ME, Baron JA, Lieberman DA, Schatzkin A, Lanza E, Winawer SJ, Zauber AG, Jiang R, Ahnen DJ, Bond JH, Church TR, Robertson DJ, Smith-Warner SA, Jacobs ET, Alberts DS, Greenberg ER. A pooled analysis of advanced colorectal neoplasia diagnoses after colonoscopic polypectomy. Gastroenterology. 2009 Mar;136(3):832-41. doi: 10.1053/j.gastro.2008.12.007. Epub 2008 Dec 9. PMID 19171141
- [Background] Cooper GS, Xu F, Barnholtz Sloan JS, Schluchter MD, Koroukian SM. Prevalence and predictors of interval colorectal cancers in medicare beneficiaries. Cancer. 2012 Jun 15;118(12):3044-52. doi: 10.1002/cncr.26602. Epub 2011 Oct 11. PMID 21989586
- [Background] Kaminski MF, Regula J, Kraszewska E, Polkowski M, Wojciechowska U, Didkowska J, Zwierko M, Rupinski M, Nowacki MP, Butruk E. Quality indicators for colonoscopy and the risk of interval cancer. N Engl J Med. 2010 May 13;362(19):1795-803. doi: 10.1056/NEJMoa0907667. PMID 20463339
- [Background] Corley DA, Levin TR, Doubeni CA. Adenoma detection rate and risk of colorectal cancer and death. N Engl J Med. 2014 Jun 26;370(26):2541. doi: 10.1056/NEJMc1405329. No abstract available. PMID 24963577
- [Background] Sawicki T, Ruszkowska M, Danielewicz A, Niedzwiedzka E, Arlukowicz T, Przybylowicz KE. A Review of Colorectal Cancer in Terms of Epidemiology, Risk Factors, Development, Symptoms and Diagnosis. Cancers (Basel). 2021 Apr 22;13(9):2025. doi: 10.3390/cancers13092025. PMID 33922197
- [Background] May FP, Shaukat A. State of the Science on Quality Indicators for Colonoscopy and How to Achieve Them. Am J Gastroenterol. 2020 Aug;115(8):1183-1190. doi: 10.14309/ajg.0000000000000622. PMID 32759620
- [Background] Shao PP, Bui A, Romero T, Jia H, Leung FW. Adenoma and Advanced Adenoma Detection Rates of Water Exchange, Endocuff, and Cap Colonoscopy: A Network Meta-Analysis with Pooled Data of Randomized Controlled Trials. Dig Dis Sci. 2021 Apr;66(4):1175-1188. doi: 10.1007/s10620-020-06324-0. Epub 2020 May 25. PMID 32451757
- [Background] Chang TL, Lewis B, Deutsch N, Nulsen B. Changes in Adenoma Detection Rate From Full-Spectrum Endoscopy to Standard Forward-Viewing Endoscopy. J Clin Gastroenterol. 2023 Apr 1;57(4):404-409. doi: 10.1097/MCG.0000000000001706. PMID 35470297
- [Background] Calcara C, Aseni P, Siau K, Gambitta P, Cadoni S. Water immersion sigmoidoscopy versus standard insufflation for colorectal cancer screening: A cohort study. Saudi J Gastroenterol. 2022 Jan-Feb;28(1):39-45. doi: 10.4103/sjg.sjg_198_21. PMID 34494603
- [Background] Kim SY, Lee SJ, Chung JW, Kwon KA, Kim KO, Kim YJ, Kim JH, Park DK. Efficacy of repeat forward-view examination of the right-sided colon during colonoscopy: A prospective randomized controlled trial. J Gastroenterol Hepatol. 2020 Oct;35(10):1746-1752. doi: 10.1111/jgh.15064. Epub 2020 Apr 20. PMID 32267568
- [Background] Rath T, Pfeifer L, Neufert C, Kremer A, Leppkes M, Hoffman A, Neurath MF, Zopf S. Retrograde inspection vs standard forward view for the detection of colorectal adenomas during colonoscopy: A back-to-back randomized clinical trial. World J Gastroenterol. 2020 Apr 28;26(16):1962-1970. doi: 10.3748/wjg.v26.i16.1962. PMID 32390706
- [Background] Kamal F, Khan MA, Lee-Smith W, Sharma S, Acharya A, Imam Z, Farooq U, Hanson J, Pulous V, Aziz M, Chandan S, Kouanda A, Dai SC, Munroe CA, Howden CW. Second exam of right colon improves adenoma detection rate: Systematic review and meta-analysis of randomized controlled trials. Endosc Int Open. 2022 Oct 17;10(10):E1391-E1398. doi: 10.1055/a-1896-4499. eCollection 2022 Oct. PMID 36262512
- [Background] Nunez Rodriguez MH, Diez Redondo P, Riu Pons F, Cimavilla M, Hernandez L, Loza A, Perez-Miranda M. Proximal retroflexion versus second forward view of the right colon during screening colonoscopy: A multicentre randomized controlled trial. United European Gastroenterol J. 2020 Jul;8(6):725-735. doi: 10.1177/2050640620924210. Epub 2020 May 7. PMID 32379535
- [Background] Desai M, Bilal M, Hamade N, Gorrepati VS, Thoguluva Chandrasekar V, Jegadeesan R, Gupta N, Bhandari P, Repici A, Hassan C, Sharma P. Increasing adenoma detection rates in the right side of the colon comparing retroflexion with a second forward view: a systematic review. Gastrointest Endosc. 2019 Mar;89(3):453-459.e3. doi: 10.1016/j.gie.2018.09.006. Epub 2018 Sep 14. PMID 30222971
- [Derived] Han F, Zhou H, Wang H, Zhang L, Ren W, Wang N, Hou Y, Deng Y, Li X, Yao J. Effect of Second Sigmoid Colon Intubation During Colonoscopy on Adenoma Detection Rate in Overweight and Obese Patients: A Prospective Randomized Controlled Trial. Am J Gastroenterol. 2025 Jun 26. doi: 10.14309/ajg.0000000000003611. Online ahead of print. PMID 40569306

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT06186778/Prot_SAP_000.pdf
  • Informed Consent Form (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/78/NCT06186778/ICF_001.pdf